CLINICAL TRIAL: NCT00239460
Title: Efficacy and Safety (Including 24-hour Holter Monitoring) of Tiotropium Inhalation Capsules in Patients With Chronic Obstructive Pulmonary Disease (a 12-week, Parallel Group, Randomized, Placebo-cotrolled, Double-blind Study).
Brief Title: Efficacy and Safety (Including 24-hour Holter Monitoring) of Tiotropium Inhalation Capsules in Patients With COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.284
Record Dates: First submitted 2005-10-14; First posted 2005-10-17 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

INTERVENTIONS:
Drug: Tiotropium

SUMMARY:
The objective of this study is to evaluate the effect of inhaled tiotropium bromide on trough FEV1 and to assess the cardiac effects through 12-lead and Holter ECG monitoring in patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* History of COPD, FEV1 less than or equal to 65%, FEV1/FVC less than or equal 70%
* Smoking history greater than or equal to 10 pack years
* Not history of clinical diagnosis of asthma and/or atopy
* A history of thoracotomy with pulmonary resection
* Patients requiring the use of supplemental oxygen therapy for >12 hours per day
* Chronic use of systemic corticosteroids in an unstable daily dose
* Patients with a recent history of myocardial infarction
* A known hypersensitivity to anticholinergic drugs

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196
Dates: Start 2003-07; Primary Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Trough FEV1 after 12 weeks of treatment | 12 weeks

SECONDARY OUTCOMES:
Trough FEV1 at Visit 3 | week 8
Trough FVC at Visits 3 and 4 | week 8 and week 12
FEV1 and FVC 90 min post study drug inhalation at all visits | 90 minutes post-medication
Use of rescue medication | 12 weeks
Patient's Global Evaluation | week 8 and week 12
Physician's Global Evaluation | week 8 and week 12
Health Related Quality of Life assessed by the EQ5D at Visit 2 and 4 | week 8 and week 12
Adverse events | 12 weeks
Vital signs | week 8 and week 12
Physical Exam | week 12
12-lead ECG | week 8 and week 12
24-hour holter ECG monitoring | week 8 and week 12

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim
Locations (12):
- United States (12):
  - Attn: William C. Bailey, M.D., Birmingham, Alabama
  - Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - Olive View UCLA Medical Center, Sylmar, California
  - Rocky Mountain Center for Clinical Research, Wheat Ridge, Colorado
  - Respiratory Diseases (111A), Bay Pines, Florida
  - Boehringer Ingelheim Investigational Site, Pembroke Pines, Florida
  - Boehringer Ingelheim Investigational Site, Coeur d'Alene, Idaho
  - LSU Health Sciences Center, Shreveport, Louisiana
  - Pulmonary and Critical Care Services, PC, Albany, New York
  - The Oregon Clinic, Portland, Oregon
  - Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - Boehringer Ingelheim Investigational Site, Houston, Texas

REFERENCES:
- [Derived] Hohlfeld JM, Furtwaengler A, Konen-Bergmann M, Wallenstein G, Walter B, Bateman ED. Cardiac safety of tiotropium in patients with COPD: a combined analysis of Holter-ECG data from four randomised clinical trials. Int J Clin Pract. 2015 Jan;69(1):72-80. doi: 10.1111/ijcp.12596. Epub 2014 Dec 11. PMID 25496316